CLINICAL TRIAL: NCT02744781
Title: Smaller Size and Asymmetry of Trunk Muscles in Combat Sports Athletes With Lumbar Intervertebral Disc Degeneration
Brief Title: Trunk Muscles and Lumbar Intervertebral Disc Degeneration in Combat Sports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Technology, Hiroshima College (Other)
Responsible Party: Principal Investigator, IWAI Kazunori, Associate Professor, National Institute of Technology, Hiroshima College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NITHiroshimaC
Record Dates: First submitted 2016-03-28; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Other Intervertebral Disc Degeneration, Lumbar Region
Keywords: Muscular Atrophy; Asymmetry; Athletes
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lumbar disc degeneration; LDD (Experimental): The LDD group included subjects with at least 1 abnormal disc from L1-2 to L5-S1 of grade III, IV, or V. The non-LDD group included subjects with 5 normal discs of grade I or II. For further assessment, the most damaged disc of the 5 constituted the highest grade of LDD.
  Interventions: Device: Lumbar disc degeneration; LDD

INTERVENTIONS:
Device: Lumbar disc degeneration; LDD — All MR images, taken at 5 lumbar intervertebral disc levels from the first lumbar (L1) vertebra to the first sacral vertebra (S1), were independently evaluated by 2 experienced orthopedic specialists in a random order using a grading system for LDD assessment. Using a comprehensive grading system for LDD, discs were classified into 5 grades, as described by Pfirrman et al. This system uses characteristics of disc structure, distinction between the nucleus and annulus, MRI signal intensity, and intervertebral disc height for grading, and has been accepted as a standardized and reliable evaluation tool for assessment of MRI disc morphology.

SUMMARY:
This study examined whether there is an association between the presence of lumbar intervertebral disc degeneration (LDD) and the size and symmetry of the cross-sectional areas (CSAs) of the trunk muscles in combat sports athletes. Participants in this study were collegiate combat sports athletes. All intervertebral discs from L1/2 to L5/S1 in all athletes were assessed using MRI and a comprehensive grading system of LDD (grades I-V). All 151 athletes were divided into 2 groups: LDD and non-LDD. CSAs of trunk muscles at the L3/4 disc level were measured on MRI.

DETAILED DESCRIPTION:
The athletes lay on a bed in the MR imaging unit in a comfortable and relaxed supine position. MR imaging was performed with a 0.3-T MR using surface coils with the body coil in the supine position (AIRIS II, Hitachi, Tokyo, Japan). T2-weighted fast spin-echo imaging was used to obtain sagittal images of the lumbar spine and intervertebral discs (repetition time, 3000 ms; echo time, 112 ms; matrix, 256 × 265; field of view, 320 mm; slice thickness, 10 mm).

All MR images, taken at 5 lumbar intervertebral disc levels from the first lumbar (L1) vertebra to the first sacral vertebra (S1), were independently evaluated by 2 experienced orthopedic specialists in a random order using a grading system for LDD assessment. Using a comprehensive grading system for LDD, discs were classified into 5 grades, as described by Pfirrman et al. This system uses characteristics of disc structure, distinction between the nucleus and annulus, MRI signal intensity, and intervertebral disc height for grading, and has been accepted as a standardized and reliable evaluation tool for assessment of MRI disc morphology. The assessment was blinded so as not to disclose any knowledge about the athlete's condition, such as the subjective functional disability level of LBP. When the 2 experienced orthopedic specialists had differing opinions on disc grades, the disagreements were debated and resolved with discussion.

The 151 participating athletes were divided into 2 groups: LDD and non-LDD. The LDD group included subjects with at least 1 abnormal disc from L1-2 to L5-S1 of grade III, IV, or V. The non-LDD group included subjects with 5 normal discs of grade I or II. For further assessment, the most damaged disc of the 5 constituted the highest grade of LDD.

CSAs of trunk muscles Transverse MR spin-echo T1-weighted images were obtained at the L3-4 level parallel to the lumbar disc space (repetition time, 760 ms; echo time, 20 ms; matrix, 256 × 265; field of view, 320 mm; slice thickness, 5.0 mm). The image was traced onto paper and the traced image was then transferred to a computer in order to measure CSAs. CSAs were calculated using image analysis software (Scion Image Beta 4.02, Scion Corp., Frederick, MD, USA), and grouped into 5 large areas because they had poorly defined borders. Each of the 5 areas was represented by the same CSA on the left and right sides of the transverse image (rectus abdominis, obliques, psoas, quadratus lumborum, and lumbar erector spinae plus multifidus). The 5 areas were summed to determine the total area. Three of the CSAs included multiple muscles: obliques, psoas, and lumbar erector spinae). Oblique muscles comprise the internal and external obliques and transversus abdominis. Psoas muscles comprise the psoas major and minor muscles. The lumbar erector spinae includes the iliocostalis, longissimus, and spinalis. All CSAs were normalized by dividing the values by the athlete's body weight. This method was used because most of the combat sports adopt the weight category system, and a previous study reported the correlation between CSAs of the trunk muscles in athletes according to their body mass.

ELIGIBILITY:
Inclusion Criteria:

* collegiate high-level combat athletes

Exclusion Criteria:

* previous lumbar surgery and specific low back pain

Ages: 19 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2001-04; Primary Completion 2004-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Cross-sectional area or trunk muscles | an average of 1 month
  Transverse MR spin-echo T1-weighted images

IPD SHARING:
Plan to Share IPD: Yes